CLINICAL TRIAL: NCT03432676
Title: Single-Arm, Phase II Proof of Concept Study of IDO-1 Inhibitor Epacadostat in Combination With Pembrolizumab in Advanced Pancreatic Cancer With Chromosomal Instability/Homologous Recombination Repair Deficiency (HRD)
Brief Title: Epacadostat and Pembrolizumab in Treating Participants With Advanced Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Incyte (supporter of the study) is no longer going to support the study.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0893; NCI-2018-00912 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0893 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-02-06; First posted 2018-02-14 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: ATM Gene Mutation; Deleterious BRCA1 Gene Mutation; Deleterious BRCA2 Gene Mutation; Homologous Recombination Deficiency; Pancreatic Ductal Adenocarcinoma; Stage II Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8; Stage IIB Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — epacadostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, epacadostat) (Experimental): Participants receive pembrolizumab IV over 30 minutes on day 1 and epacadostat PO BID on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Epacadostat; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Epacadostat — Given PO
  Other Names: INCB 024360; INCB024360
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well epacadostat and pembrolizumab work in treating participants with pancreatic cancer that has spread to other places in the body. Epacadostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving epacadostat and pembrolizumab may work better in treating participants with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of epacadostat in combination with pembrolizumab as determined by the best overall response rate in previously treated patients with advanced pancreatic adenocarcinoma with homologous recombination repair deficiency (HRD) aberrations.

SECONDARY OBJECTIVES:

I. To further determine the efficacy of epacadostat in combination with pembrolizumab in previously treated patients with advanced pancreatic adenocarcinoma with HRD aberrations.

II. To assess the safety and tolerability of epacadostat in combination with pembrolizumab in previously treated patients with advanced pancreatic adenocarcinoma with HRD aberrations.

EXPLORATORY OBJECTIVES:

I. To identify predictive, mechanistic, and/or surrogate biomarkers of clinical efficacy of epacadostat in combination with pembrolizumab in previously treated patients with advanced pancreatic adenocarcinoma with HRD aberrations utilizing exploratory studies investigating the patients tumor and immune system response including: flow cytometry of fresh peripheral blood mononuclear cell (PBMC), PDL-1.

OUTLINE:

Participants receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and epacadostat orally (PO) twice daily (BID) on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, participants are followed up at 30 days, every 8 weeks for 3 years, and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Have received at least one prior therapy for metastatic disease
* Patients with HRD identified by one of the following criteria: a) Tested positive for BRCA 1 or 2 germline deleterious mutation, b) Previously identified genetic aberrations that are associated with HRD (e.g., somatic BRCA mutation, PALB2, Fanconi anemia gene or RAD51 mutations), c) Patients with somatic ATM loss as identifiable with immunohistochemistry or with ATM mutation, d) Pancreatic ductal adenocarcinoma (PDAC) patients with family history of 2 or more first-degree relatives with BRCA-associated cancers (stomach, breast, ovary) or 1 or more first-degree relative with PDAC
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or at least one site of disease must be uni-dimensionally measurable as per RECIST 1.1. All radiology studies must be performed within 28 days prior to registration
* Patients must have an archival sample of tumor or metastatic site core biopsy to be eligible
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Within 10 days of treatment initiation: Absolute neutrophil count (ANC) >= 1.5 x 109/L
* Within 10 days of treatment initiation: platelet count >= 100 x 109/L
* Within 10 days of treatment initiation: hemoglobin >= 9 g/dl without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Within 10 days of treatment initiation: If serum creatinine concentration >= 1.5 x upper limit of normal (ULN), then estimated creatinine clearance must be >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN
* Within 10 days of treatment initiation: total bilirubin =< 1.5 x ULN (3 x ULN if a exists a history of Gilbert syndrome) or direct bilirubin >= ULN for subjects with total bilirubin levels > 1.5 ULN
* Within 10 days of treatment initiation: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN
* Within 10 days of treatment initiation: albumin >= 3 mg/dL. Creatinine clearance should be calculated per institutional standard
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects of childbearing potential must agree to use an adequate method of contraception. Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* For screening electrocardiographs (ECGs), exclude patients with a Fridericia's corrected QT interval (QTcF) > 480 ms, or JTc > 340 ms for those with an intraventricular conduction delay. If the screening ECG has a QTcF > 480 ms, eligibility can be confirmed if the average of 3 ECGs done 5 minutes apart have an average QTcF < 480 ms
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or epacadostat or any of their excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-IDO-1 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy
* Has ascites that requires frequent paracentesis or a pleural effusion that requires repeated thoracentesis
* Has arterial vascular involvement
* Has received monoamine oxidase inhibitors within 21 days prior to starting study
* Has any history of serotonin syndrome after receiving serotonergic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-31 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Best objective response rate | Up to 2 years
  The objective response rate (partial response [PR] + complete response [CR]) and its corresponding exact 1-sided 90% confidence interval (CI) will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Milind Javle, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org